CLINICAL TRIAL: NCT01348048
Title: Danish Palliative Care Trial (DanPaCT): A Randomised Clinical Multi-centre Trial Investigating the Effect of Specialised Palliative Care on Symptoms, Survival, Economical Factors and Satisfaction in Patients With Cancer Reporting Palliative Needs
Brief Title: A Trial Investigating the Effect of Specialised Palliative Care on Symptoms, Survival, Economical Factors and Satisfaction
Acronym: DanPaCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: TRYG Foundation (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Mogens Groenvold, MD, PhD, DMSc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DanPaCT2011
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Cancer
Keywords: palliative care; end-of-life care; randomized clinical trial; quality of life; needs assessment; patient satisfaction; cost-effectiveness; Screening
MeSH Terms: conditions — Neoplasm Metastasis; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialised palliative care (SPC) group (Experimental): Patients continue with their standard treatment (typically they receive treatment in one or more hospitals departments and from their GP). In addition, they are offered a consultation in the SPC out-patient clinic (or at home if the patient cannot attend the hospital) as soon as possible and no more than one week after randomization. If possible, each patient will have at least two contacts to the SPC in the trial period.
  Interventions: Other: Specialised palliative care (SPC)
- Standard care group (No Intervention): Patients continue with their standard treatment. They are instructed to contact either their GP or their hospital department if they feel that additional treatment or care is needed.

INTERVENTIONS:
Other: Specialised palliative care (SPC) — The interventions given by the SPC centres follow the the WHO and the EAPC guidelines for palliative care. It is not possible in advance to describe the interventions more specifically as these will be adjusted to each particular patient. As part of the study the medical records of all patients in the intervention group will be reviewed with the purpose of describing the interventions given for the different symptoms and problems.
  Arms: Specialised palliative care (SPC) group

SUMMARY:
Specialised palliative care (SPC) seeks to relieve suffering and improve quality of life in patients with a life threatening disease such as advanced cancer. Many patients with advanced cancer are not in contact with SPC. Previous studies have shown that among advanced cancer patients not referred to SPC there is a significant prevalence of symptoms, problems and needs. The aims of the present study are to investigate whether patients with metastatic cancer, who report palliative needs in a screening, will benefit from being referred to SPC and to investigate the economical consequences of such a referral.

DETAILED DESCRIPTION:
The trial is a randomised, clinical, multicenter trial including 6 Danish SPC-centres. The basic principle is that patients with palliative needs (see inclusion criteria) are identified at oncological departments and randomised to either (i) standard treatment plus SPC (intervention group) or (ii) standard treatment (control group).

Patients will be identified by the following procedure: A) Each week a research nurse reviews the medical records of consecutive patients seen in oncological out-patients clinic. B) Eligible patients are asked to fill out a questionnaire (the screening) that investigates symptoms and problems. The patients are told that their questionnaire will be evaluated and that the research nurse will contact some of the patients later on with information about a RCT. C) Those patients who report at least one palliative need in the questionnaire (see inclusion criteria) and have four additional symptoms are contacted by the research nurse who provide the patients with written and verbal information about the RCT. D) Patients who give informed consent are randomised.

Detailed statistical analysis plan:

Analysis of the primary outcome The primary outcome analysis will be a modified ITT analysis. Patients who withdrew consent after randomisation, who were randomised by mistake and did not fulfil our inclusion criteria, or who were not alive at the time of the follow-ups, will be excluded from the primary analysis. All exclusions will be shown in the CONSORT flow-chart of patient participation.

In the primary outcome analysis we will use multiple imputation for non-responders if there are more than 5% missing outcomes. In total, we will make 20 different data-sets with imputation based on a regression model using predictive-mean-matching using the MI and the MI ANALYSIS procedures in SAS. The primary outcome analysis will be made as a multiple regressions adjusted for the stratification variable if it is normally distributed.

Sensitivity analyses of the primary outcome We will make five sensitivity analyses: 1) a fully adjusted analysis including all relevant covariates, 2) a complete case analysis, 3) an analysis including a model for repeated measurement, 4) a per protocol analysis, 5) an analysis including imputations for those who died.

Analysis of secondary outcomes The analyses of the seven scales from EORTC QLQ-C30 (physical function, role function, emotional function, nausea and vomiting, pain, dyspnoea, or lack of appetite) will be made using the same principles as described for the primary outcome including the sensitivity analyses. Survival will be analysed using Kaplan-Meier plot. Patients who are alive three months after the end of data-collection will be censured on this date. A Cox regression will be made adjusted for the stratification variable. A sensitivity analysis will be made adjusting for all relevant covariates.

Exploratory outcomes and subgroup analyses For serious adverse events we report the number of hospitalisations, the number of acute hospitalisations and the number of deaths in the eight week trial period. The analyses of the other exploratory outcomes will not be dealt with in detail here. The overall principles regarding questionnaire data (the remaining scales from EORTC QLQ-C30, HADS and FAMCARE-P16) are that they will be analysed as complete case analyses.

Significance levels All tests will be two-tailed. For the primary outcome the risk of type I error is set to 5% (i.e., a significance level of P<0.05). As we have 8 secondary outcomes, we adjust the significance levels to P<0.01 to control the familywise (or cumulative) type I error due to multiplicity. The P-values of the exploratory outcomes will be provided, but it will be made clear that the analyses are exploratory.

Register-data, data-management and analyses Survival will be retrieved from the Danish Civil Registration System (CPR), and serious adverse events and contacts from The Danish Patient Registry (Landspatientregistret).

Data management will be done by project manager Anna Thit Johnsen. Analyses will be made by statistician Morten Aa. Petersen, who is blinded to the identity of the two intervention groups, which will be denoted Y and X. Results will be presented blinded in the same way for the investigators, and conclusions regarding the results will be drawn by the investigators and written down while the interventions are still blinded. The blinding will not be broken before all analyses of primary and secondary outcomes have been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Cancer stage 4 according to the TNM system (for patients with cancer in CNS inclusion criteria is: cancer grade three or four and no possibility of radical treatment)
* At least 18 years
* Live in the area of the participating hospitals
* No contact with specialised palliative care within the previous year
* At least one palliative need defined as a EORTC QLQ-C30 scale score of at least 50% of the score corresponding to maximal symptomatology or maximal functional impairment
* Four additional symptoms (defined as patients answering, on average, at least 'a little' in any of the 14 function or symptom scales in the EORTC QLQ-C30 questionnaire)
* Written informed consent

Exclusion Criteria:

* Do not understand Danish well enough to participate in the study
* Are judged incapable of co-operating with the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the EORTC QLQ-C30 scale that constitutes the patient's primary need | Baseline, 3 weeks and 8 weeks
  The difference between the intervention and the control group in the change from baseline to the weighted mean of the 3- and 8-week follow-up (measured as AUC) for the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scale score that constitutes the primary need. The primary need can be a need related to the following: physical function, role function, emotional function, pain, shortness of breath, lack of appetite and nausea/vomiting.

SECONDARY OUTCOMES:
Patients reported symptoms and problems according to the EORTC QLQ-C30 | Baseline, 3 weeks and 8 weeks
  The difference between the intervention and the control group in the change from baseline to the weighted mean of the 3- and 8-week follow-up (measured as AUC) for all the symptoms and problems measured by the EORTC QLQ-C30 and for anxiety and depression measured by the The Hospital Anxiety and Depression Scale (HAD scale)
Survival | From the start of the trial to minimum three months after the end of the intervention.
  Survival.
Economical consequences | From the start of the trial to minimum three months after the end of the intervention.
  Economical consequences measured as the expenses to health care services (treatments, hospitalisation, outpatient visits, emergency room visits, and visits with the general practitioner).
Patient reported Satisfaction with services provided by the health care system measured with the questionnaire FAMCARE-p16 | 8 weeks
  The difference between the intervention and the control group in the change from baseline to the weighted mean of the 3- and 8-week follow-up (measured as AUC) in the patients' evaluation of treatment and care provided by the health care system measured by the FAMCARE-p16 and four additional items developed for this trial

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Groenvold, MD, PhD, DMSc, Principal Investigator — Department of Palliative Medicine, Bispebjerg Hospital
Locations (6):
- Denmark (6):
  - The Palliative Team, Aarhus University Hospital, Aarhus
  - Section of Acute Pain Management and Palliative Medicine, Rigshospitalet, Copenhagen
  - Department of Palliative Medicine, Bispebjerg Hospital, Copenhagen
  - Palliative Team Herning, Herning
  - Palliative Team Fyn, Odense University hospital, Nyborg
  - Palliative Team Vejle, Vejle

REFERENCES:
- [Background] Johnsen AT, Damkier A, Vejlgaard TB, Lindschou J, Sjogren P, Gluud C, Neergaard MA, Petersen MA, Lundorff LE, Pedersen L, Fayers P, Stromgren AS, Higginson IJ, Groenvold M. A randomised, multicentre clinical trial of specialised palliative care plus standard treatment versus standard treatment alone for cancer patients with palliative care needs: the Danish palliative care trial (DanPaCT) protocol. BMC Palliat Care. 2013 Oct 24;12(1):37. doi: 10.1186/1472-684X-12-37. PMID 24152880
- [Background] Johnsen AT, Petersen MA, Gluud C, Lindschou J, Fayers P, Sjogren P, Pedersen L, Neergaard MA, Vejlgaard TB, Damkier A, Nielsen JB, Stromgren AS, Higginson IJ, Groenvold M. Detailed statistical analysis plan for the Danish Palliative Care Trial (DanPaCT). Trials. 2014 Sep 26;15:376. doi: 10.1186/1745-6215-15-376. PMID 25257804
- [Derived] Skjoedt N, Johnsen AT, Sjogren P, Neergaard MA, Damkier A, Gluud C, Lindschou J, Fayers P, Higginson IJ, Stromgren AS, Groenvold M. Early specialised palliative care: interventions, symptoms, problems. BMJ Support Palliat Care. 2021 Dec;11(4):444-453. doi: 10.1136/bmjspcare-2019-002043. Epub 2020 Mar 27. PMID 32220944
- [Derived] Johnsen AT, Petersen MA, Sjogren P, Pedersen L, Neergaard MA, Damkier A, Gluud C, Fayers P, Lindschou J, Stromgren AS, Nielsen JB, Higginson IJ, Groenvold M. Exploratory analyses of the Danish Palliative Care Trial (DanPaCT): a randomized trial of early specialized palliative care plus standard care versus standard care in advanced cancer patients. Support Care Cancer. 2020 May;28(5):2145-2155. doi: 10.1007/s00520-019-05021-7. Epub 2019 Aug 13. PMID 31410598
- [Derived] Groenvold M, Petersen MA, Damkier A, Neergaard MA, Nielsen JB, Pedersen L, Sjogren P, Stromgren AS, Vejlgaard TB, Gluud C, Lindschou J, Fayers P, Higginson IJ, Johnsen AT. Randomised clinical trial of early specialist palliative care plus standard care versus standard care alone in patients with advanced cancer: The Danish Palliative Care Trial. Palliat Med. 2017 Oct;31(9):814-824. doi: 10.1177/0269216317705100. Epub 2017 May 12. PMID 28494643